CLINICAL TRIAL: NCT05033184
Title: Effectiveness of a Brief Internet-delivered Behaviour Change Intervention Among Healthy Middle-aged Adults: A Randomized Controlled Trial
Brief Title: Effectiveness of a Brief Internet-delivered Behaviour Change Intervention Among Healthy Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-074
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2022-11

CONDITIONS: Health Behavior
Keywords: Physical Activity; Control Beliefs; Emotion Regulation; Resilience; Social Support
MeSH Terms: conditions — Health Behavior; Motor Activity; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Action Planning Exercise (Experimental)
  Interventions: Behavioral: Brief Action Planning Exercise
- Goal Setting Exercise (Active Comparator)
  Interventions: Behavioral: Goal Setting Exercise

INTERVENTIONS:
Behavioral: Brief Action Planning Exercise — The Brief Action Planning exercise is a previously developed goal-setting exercise which has been designed to incorporate aspects of motivational interviewing such as compassion, acceptance, evocation, and partnership. It is a tool that allows participants to identify an aspect of their life they would like to improve upon and guides them through the process of making a specific, measurable, achievable, realistic, and timely (SMART) goal. It also assesses their confidence in achieving this goal so as to assist with making alternative plans if confidence is low.
  Arms: Brief Action Planning Exercise
Behavioral: Goal Setting Exercise — The Goal Setting exercise allows participants to identify an aspect of their life they would like to improve upon without incorporating aspects of motivational interviewing components or providing any guidance on how to set this goal.
  Arms: Goal Setting Exercise

SUMMARY:
Previous studies have demonstrated the need to move beyond the common misconception of midlife as a time of crisis so that further understandings of the midlife as a time of opportunity for the maintenance and improvement of health can be developed. Several psychosocial factors such as resilience, emotion regulation, perceived social support, and control beliefs have been identified as having a role in the adoption of healthier lifestyle habits in middle age which, in turn, may decrease the risk of a developing or worsening chronic disease. Several behaviour change interventions have also been proposed in the literature. As Canada's population ages, it is important that brief behaviour change interventions, and the psychosocial factors that facilitate such behaviour changes, be identified as a way to promote better health during the midlife years so as to improve the experience of aging. The present study is aimed at evaluating the influence of psychosocial factors on the adoption of healthy lifestyle habits. Specifically, this study aims to examine whether differing experiences of social support, resilience, emotion regulation, and control beliefs influence physical activity levels following a brief behaviour change intervention. Participants will be asked to complete a demographics questionnaire followed by a series of measures to determine the individual's perceived levels of social support, resilience, emotion regulation, and control beliefs. After completing this set of questionnaires, participants will be randomly assigned to either an experimental or a control condition. Participants in the experimental condition will be asked to complete the Brief Action Planning exercise as a way to identify a goal related to health behaviours. Participants in the control condition will be asked to identify a goal related to health behaviours without being introduced to the Brief Action Planning exercise. Two weeks and four weeks following this intervention, individuals will be asked to indicate the degree to which they were able to achieve their health goal. It is expected that individuals in the experimental condition will experience greater improvement in physical activity levels compared to individuals in the control condition. The investigators also anticipate that improvements in physical activity levels in the experimental condition will be influenced by the psychosocial factors of social support, resilience, emotion regulation, and control beliefs. The potential significance of this study includes increasing awareness of the influence of psychosocial factors on health behaviours and the possible effectiveness of a brief behaviour change intervention among middle-aged adults. Potential interventions may be used in clinical settings or community programs in which middle-aged adults engage.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Saskatchewan, Canada
* Between the ages of 35 and 64 years
* Deemed eligible to increase physical activity levels by the Physical Activity Readiness Questionnaire for Everyone (Par-Q+; Canadian Society for Exercise Physiology, 2019)

Exclusion Criteria:

* Residing outside of Saskatchewan, Canada
* Under the age of 35 years or over the age of 64 years
* Deemed ineligible to increase physical activity levels by the Physical Activity Readiness Questionnaire for Everyone (Par-Q+; Canadian Society for Exercise Physiology, 2019)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (Baseline) | Baseline Period
  Our final outcome measure will be the International Physical Activity Questionnaire (IPAQ). The IPAQ will measure the degree to which participants spent time on vigorous, moderate, walking, and sitting activities. The IPAQ gets scored as categories (low activity levels, moderate activity levels, and high activity levels). A score of high activity levels is assigned to those who engage in vigorous activities at least 3 days a week OR 7 or more days of any combination of walking, moderate intensity, or vigorous activities. A score of moderate levels of physical activity will be assigned to those who engage in 3 or more days of vigorous activity and/ or walking of at least 30 minutes per day OR 5 or more days of moderate intensity activity and/or walking at least 30 minutes per day OR 5 or more days of any combination of walking, moderate intensity or vigorous activities. Those who do not meet the criteria for either vigorous or moderate will be scored as having low levels of activity.
International Physical Activity Questionnaire (Follow-Up 1) | 2-Week Follow-Up Period
  Our final outcome measure will be the International Physical Activity Questionnaire (IPAQ). The IPAQ will measure the degree to which participants spent time on vigorous, moderate, walking, and sitting activities. The IPAQ gets scored as categories (low activity levels, moderate activity levels, and high activity levels). A score of high activity levels is assigned to those who engage in vigorous activities at least 3 days a week OR 7 or more days of any combination of walking, moderate intensity, or vigorous activities. A score of moderate levels of physical activity will be assigned to those who engage in 3 or more days of vigorous activity and/ or walking of at least 30 minutes per day OR 5 or more days of moderate intensity activity and/or walking at least 30 minutes per day OR 5 or more days of any combination of walking, moderate intensity or vigorous activities. Those who do not meet the criteria for either vigorous or moderate will be scored as having low levels of activity.
International Physical Activity Questionnaire (Follow-Up 2) | 4-Week Follow-Up Period
  Our final outcome measure will be the International Physical Activity Questionnaire (IPAQ). The IPAQ will measure the degree to which participants spent time on vigorous, moderate, walking, and sitting activities. The IPAQ gets scored as categories (low activity levels, moderate activity levels, and high activity levels). A score of high activity levels is assigned to those who engage in vigorous activities at least 3 days a week OR 7 or more days of any combination of walking, moderate intensity, or vigorous activities. A score of moderate levels of physical activity will be assigned to those who engage in 3 or more days of vigorous activity and/ or walking of at least 30 minutes per day OR 5 or more days of moderate intensity activity and/or walking at least 30 minutes per day OR 5 or more days of any combination of walking, moderate intensity or vigorous activities. Those who do not meet the criteria for either vigorous or moderate will be scored as having low levels of activity.

SECONDARY OUTCOMES:
Confidence (Baseline) | Baseline Period
  The Confidence outcome asks the participant to rate how confident they feel in following their plan The degree to which participants report that they are confident about carrying out their plan over the next two weeks on a scale from 1 to 10, with scores above 7 indicating high confidence and scores below 7 indicating low confidence.
Confidence (Follow-Up) | 2-Week Follow-Up Period
  The Confidence outcome asks the participant to rate how confident they feel in following their plan The degree to which participants report that they are confident about carrying out their plan over the next two weeks on a scale from 1 to 10, with scores above 7 indicating high confidence and scores below 7 indicating low confidence.
Achievement (Follow-Up 1) | 2-Week Fellow-Up Period
  The Achievement outcome asks the participant to rate the degree to which they followed their plan over the previous two weeks by selecting either 'fully,' 'partially,' or 'not at all.'
Achievement (Follow-Up 2) | 4-Week Follow-Up Period
  The Achievement outcome asks the participant to rate the degree to which they followed their plan over the previous two weeks by selecting either 'fully,' 'partially,' or 'not at all.'

CONTACTS AND LOCATIONS:
Overall Officials: Natasha L Gallant, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
The study's principal investigator, supervisor, and project investigators will be the only persons with access to the data.

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Warburton DER, Jamnik VK, Bredin SSD, Gledhill N on behalf of the PAR-Q+ Collaboration. The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and Electronic Physical Activity Readiness Medical Examination (ePARmed-X+). Health & Fitness Journal of Canada. 2011; 4(2): 3-23.
- [Background] Infurna FJ, Gerstorf D, Lachman ME. Midlife in the 2020s: Opportunities and challenges. Am Psychol. 2020 May-Jun;75(4):470-485. doi: 10.1037/amp0000591. PMID 32378943
- [Background] Lachman ME, Teshale S, Agrigoroaei S. Midlife as a Pivotal Period in the Life Course: Balancing Growth and Decline at the Crossroads of Youth and Old Age. Int J Behav Dev. 2015 Jan 1;39(1):20-31. doi: 10.1177/0165025414533223. PMID 25580043
- [Background] Gutnick D, Reims K, Davis C, Gainforth H, Jay M, Cole S. Brief action planning to facilitate behavior change and support patient self-management. Journal of Clinical Outcomes Management. 2014; (21)1: 17-29.